CLINICAL TRIAL: NCT00070317
Title: Lymphatic Mapping and Sentinel Node Identification in Patients With Stage1B1 Cervical Carcinoma
Brief Title: Lymph Node Mapping and Sentinel Lymph Node Identification in Patients With Stage IB1 Cervical Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GOG-0206; NCI-2012-02559 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000331918; GOG-0206 (Other: Gynecologic Oncology Group); GOG-0206 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2015-06

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma; Stage I Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — iso-sulfan blue; sulfan blue; Methylene Blue; Sentinel Lymph Node Biopsy; Technetium Tc 99m Sulfur Colloid

ARMS (1):
- Diagnostic (Experimental): Patients receive radiolabeled technetium Tc 99m sulfur colloid injected around the tumor 6 hours prior to or after induction of anesthesia right before surgery. Patients then undergo radical hysterectomy and complete pelvic and low para-aortic lymphadenectomy. Intraoperatively, patients undergo lymphatic mapping and sentinel lymph node identification using isosulfan blue or methylene blue injected at 4 locations in the cervix and a hand-held gamma counter.
  Interventions: Drug: Isosulfan Blue; Procedure: Lymph Node Mapping; Procedure: Lymphangiography; Drug: Methylene Blue; Procedure: Radionuclide Imaging; Procedure: Sentinel Lymph Node Biopsy; Radiation: Technetium Tc-99m Sulfur Colloid; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Isosulfan Blue — Undergo lymphangiography using isosulfan blue or methylene blue
  Other Names: Lymphazurin; N-[4-[(4-(diethylamino)phenyl)(2,5-disulfophenyl)methylene]-2,5-cyclohexadien-1-ylidene]-N-ethyl-ethanaminium hydroxide
Procedure: Lymph Node Mapping — Undergo lymphatic mapping
  Other Names: lymphatic mapping
Procedure: Lymphangiography — Undergo lymphangiography using isosulfan blue or methylene blue
  Other Names: Lymphography
Drug: Methylene Blue — Undergo lymphangiography using isosulfan blue or methylene blue
  Other Names: Azul de Metileno; Azul Metile; Blu di Metilene; CI Basic Blue 9; CI-52015; Collubleu; Colour Index No. 52015; Desmoidpillen; Methylenum Caeruleum; Methylthioninii Chloridum; Methylthioninium Chloride; Schultz No. 1038; Tetramethylthionine Chloride Trihydrate; Urolene Blue; Vitableu
Procedure: Radionuclide Imaging — Undergo radionuclide imaging with technetium Tc 99m sulfur colloid
  Other Names: nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; SCINTIGRAPHY
Procedure: Sentinel Lymph Node Biopsy — Undergo complete pelvic and low para-aortic lymphadenectomy
  Other Names: Sentinel Node Biopsy; Sentinel node biopsy alone; SLNB; SNB
Radiation: Technetium Tc-99m Sulfur Colloid — Undergo radionuclide imaging with technetium Tc 99m sulfur colloid
  Other Names: Tc 99m Sulfur Colloid; Tc-99m SC; Technetium Tc 99m Sulfur Colloid
Procedure: Therapeutic Conventional Surgery — Undergo radical hysterectomy

SUMMARY:
This clinical trial is studying how well lymph node mapping and sentinel lymph node identification work in finding lymph node metastases in patients with stage IB1 cervical cancer. Diagnostic procedures, such as lymph node mapping and sentinel lymph node identification, performed before and during surgery, may improve the ability to detect lymph node metastases in patients who have cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the sensitivity of the sentinel lymph node in the determination of lymph node metastases, using preoperative or intraoperative lymphatic mapping, in patients with stage IB1 cervical cancer.

II. Determine the false-negative predictive value of the sentinel lymph node in the determination of lymph node metastases in these patients.

OUTLINE: This is a multicenter study.

Patients receive radiolabeled technetium Tc 99m sulfur colloid injected around the tumor 6 hours prior to or after induction of anesthesia right before surgery. Patients then undergo radical hysterectomy and complete pelvic and low para-aortic lymphadenectomy. Intraoperatively, patients undergo lymphatic mapping and sentinel lymph node identification using isosulfan blue or methylene blue injected at 4 locations in the cervix and a hand-held gamma counter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of carcinoma of the cervix of 1 of the following cellular types:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Adenosquamous cell carcinoma
* Stage IB1 disease (no greater than 4 cm)
* No unequivocal evidence of metastases
* Adequate surgical candidate
* No known allergy to triphenylmethane compounds
* No prior pelvic irradiation
* No prior retroperitoneal surgery
* More than 4 weeks since prior cold knife or loop electrosurgical excision procedure (LEEP) cone biopsy
* Prior cone biopsy allowed provided current disease is stage IB1

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2004-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Levenback, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was opened to patient entry on June 21, 2004 and was closed to entry July 21, 2008.
Groups:
- Radionuclide and Isosulfan Blue Injection: Patients receive radiolabeled technetium Tc 99m sulfur colloid injected around the tumor 6 hours prior to or after induction of anesthesia right before surgery. Patients then undergo radical hysterectomy and complete pelvic and low para-aortic lymphadenectomy. Intraoperatively, patients undergo lymphatic mapping and sentinel lymph node identification using isosulfan blue or methylene blue injected at 4 locations in the cervix and a hand-held gamma counter.
  Isosulfan Blue: Undergo lymphangiography using isosulfan blue or methylene blue Lymph Node Mapping: Undergo lymphatic mapping Lymphangiography: Undergo lymphangiography using isosulfan blue or methylene blue Methylene Blue: Undergo lymphangiography using isosulfan blue or methylene blue Radionuclide Imaging: Undergo radionuclide imaging with technetium Tc 99m sulfur colloid Sentinel Lymph Node Biopsy: Undergo complete pelvic and low para-aortic lymphadenectomy Technetium Tc-99m Sulfur Colloid: Undergo radionuclid
Period: Overall Study
Arm/Group | Radionuclide and Isosulfan Blue Injection
Started | 102
Completed | 89
Not Completed | 13
Not completed — Inevaluable (Never Treated) | 1
Not completed — Ineligible Wrong Cell type/primary/stage | 3
Not completed — Ineligible required test not done | 1
Not completed — Ineligible-Improper prior treatment | 2
Not completed — Ineligible-Inadequate pathology | 6

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable patients
Groups:
- Diagnostic: Patients receive radiolabeled technetium Tc 99m sulfur colloid injected around the tumor 6 hours prior to or after induction of anesthesia right before surgery. Patients then undergo radical hysterectomy and complete pelvic and low para-aortic lymphadenectomy. Intraoperatively, patients undergo lymphatic mapping and sentinel lymph node identification using isosulfan blue or methylene blue injected at 4 locations in the cervix and a hand-held gamma counter.
  Isosulfan Blue: Undergo lymphangiography using isosulfan blue or methylene blue Lymph Node Mapping: Undergo lymphatic mapping Lymphangiography: Undergo lymphangiography using isosulfan blue or methylene blue Methylene Blue: Undergo lymphangiography using isosulfan blue or methylene blue Radionuclide Imaging: Undergo radionuclide imaging with technetium Tc 99m sulfur colloid Sentinel Lymph Node Biopsy: Undergo complete pelvic and low para-aortic lymphadenectomy Technetium Tc-99m Sulfur Colloid: Undergo radionuclid
Arm/Group | Diagnostic
Number analyzed (Participants) | 89
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 6
  30-39 years | 23
  40-49 years | 31
  50-59 years | 17
  60-69 years | 9
  70-79 years | 2
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 75
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: Sensitivity is defined as the proportion of patients who test as positive sentinel node among the patients who have lymph node metastases.
Time Frame: At the time of surgery
Population: Eligible and evaluable patients with lymph node metastasis and identified sentinel node
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Diagnostic
Number analyzed (Participants) | 21
Percentage of participants | 85.7 [67 to 96]

2. Primary Outcome: False Negative Predictive Value (FNPV)
Description: The proportion of patients with FNPV among patients who tests as negative sentinel node, where FNPV is defined as a person who tests as negative sentinel node but who actually has lymph node metastases
Time Frame: At the time of Surgery
Population: Eligible and evaluable patients who tested as negative sentinel node and have lymph node sampling
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Diagnostic
Number analyzed (Participants) | 51
Percentage of participants | 5.9 [2 to 15]

ADVERSE EVENTS:
Time Frame: All treatment-related adverse events which occurred within 30 days of study surgical procedure are reported.
Arm/Group | Diagnostic
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 0/89
Other Adverse Events (participants affected / at risk) | 32/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diagnostic (N=89)
Hemoglobin (Blood and lymphatic system disorders) | 20
Other Blood/Bone Marrow (Blood and lymphatic system disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 1
Cardiac (Cardiac disorders) | 1
Constitutional Symptoms (General disorders) | 8
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Other Gastrointestinal (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Infection (Infections and infestations) | 4
Lymphocele (Blood and lymphatic system disorders) | 1
Other Lymphatics (Blood and lymphatic system disorders) | 1
Metabolic/Laboratory (Metabolism and nutrition disorders) | 2
Pain (General disorders) | 6
Renal/Genitourinary (Renal and urinary disorders) | 3
Intra-Op Injury: Ureter (Surgical and medical procedures) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less